CLINICAL TRIAL: NCT01082510
Title: Study of the Efficacy of Maintenance Therapy by UFT or BCG for Superficial Bladder Cancer Against Recurrence in Urological Oncology Council of Northern Tokyo: EMBARK Study
Brief Title: Study of the Efficacy of Maintenance Therapy Using Uracil-tegafur (UFT) or Bacille Calmette-Guerin (BCG) for the Prevention of Recurrences of Superficial Bladder Cancer (EMBARK Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Urological Oncology Council of Northern Tokyo (Other)
Responsible Party: Shigeo Horie, Department of Urology, Teikyo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMBARK
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2010-10

CONDITIONS: Bladder Cancer
Keywords: UFT; BCG
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCG maintenance therapy (Active Comparator)
  Interventions: Drug: Bacille Calmette-Guerin
- UFT maintenance therapy (Experimental)
  Interventions: Drug: uracil-tegafur

INTERVENTIONS:
Drug: Bacille Calmette-Guerin — The patients in the BCG maintenance therapy arm will be treated with 3 successive weekly intravesical administrations of BCG at 3, 6, 12 and 18 months after the start of BCG induction therapy. The dosage of BCG used for the BCG maintenance therapy will be the same as that used for BCG induction therapy.
  Arms: BCG maintenance therapy
Drug: uracil-tegafur — The UFT maintenance therapy arm patients will be treated with the oral administration of 400 mg of UFT everyday for three years after the end of BCG induction therapy.
  Arms: UFT maintenance therapy

SUMMARY:
The purpose of this prospective randomized controlled study is to prove the non-inferiority of UFT maintenance therapy to BCG maintenance therapy for preventing recurrences of superficial bladder cancer.

DETAILED DESCRIPTION:
Patients who have undergone transurethral resection of a superficial bladder tumor (TUR-Bt) and BCG induction therapy are eligible for enrollment in this study. In principle, BCG induction therapy consists of the successive weekly intravesical administration of 81 mg of BCG-Connaught strain or 80 mg of BCG-Japan strain for 6 weeks after the completion of TUR-Bt.

The patients will be randomly assigned to a BCG maintenance therapy arm or a UFT maintenance therapy arm. The patients in the BCG maintenance therapy arm will be treated with 3 successive weekly intravesical administrations of BCG at 3, 6, 12 and 18 months after the start of BCG induction therapy. The dosage of BCG used for BCG maintenance therapy will be the same as that used for BCG induction therapy. Patients in the UFT maintenance therapy arm will be treated with the oral administration of 400 mg of UFT everyday for three years after the end of BCG induction therapy.

The primary endpoint of this study is the three-year relapse-free survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Superficial bladder cancer
* Completion of transurethral resection of bladder tumor (TUR-Bt)
* Completion of BCG induction therapy after TUR-Bt. In principle, BCG induction therapy consists of the successive weekly intravesical administration of 81 mg of BCG-Connaught strain or 80 mg of BCG-Japan strain for 6 weeks after the completion of TUR-Bt.
* Age 20 to 80 years
* ECOG performance status of 0 or 1
* Bladder capacity ≥ 150 mL
* Capable of oral UFT administration
* Expected life prognosis ≥ 3 years
* Hematopoietic WBC ≥ 3,000/mm^3
* Neutrophil ≥ 1,500/mm^3
* Platelet ≥ 100,000/mm^3
* Hepatic AST and ALT ≤ 2 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL
* Hemoglobin ≤ 9.0 g/dL
* Creatinine ≤ 1.5 mg/dL

Exclusion Criteria:

* Bladder cancer located in prostatic part of the urethra
* Anamnesis of bladder cancer classified as cT2, cT3 or cT4
* Anamnesis of metastatic bladder cancer
* Anamnesis of upper urinary tract carcinoma in situ
* Anamnestic treatment of intravesical BCG administration within previous 6 months
* Prior anticancer chemotherapy or radiotherapy
* Severe complication
* Presence of contraindications for the administration of BCG or UFT
* Pregnancy, lactation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival rate | Three-year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Teikyo University Hospital, Itabashi-ku, Tokyo, Japan